CLINICAL TRIAL: NCT03088423
Title: Tumor Response Assessment by MRI Following Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma
Brief Title: HCC Response Assessment by MRI After SBRT
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_ICL_0001
Record Dates: First submitted 2017-03-16; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: MRI; Stereotactic body radiation therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: SBRT delivers high dose selective irradiation with millimeter precision to a small volume. The Cyberknife® is a robotic SBRT dedicated device that can deliver 100 to 200 photobeams to the target — Seven to ten days before the scheduled CT, 2-4 fiducial markers were implanted percutaneously 2 to 5 cm next to the lesion under sonographic guidance following administration of local anesthesia, thus allowing real-time tracking during treatment. The total dose delivered was 45 Gy on the 80% isodose, in three fractions over 10 days. Gross tumor volume (GTV) was defined as the tumor mass that could be discerned by diagnostic imaging. An isotropic margin of 5 mm was added to account for the microscopic extension (clinical target volume, CTV) and another 3 mm margin was added to compensate for uncertainties regarding the position (previsional target volume, PTV)

SUMMARY:
The aim of this work was to describe SBRT different presentations, to study predictive factors for tumor responses following treatment, and to compare tumor response assessments according to the Response Evaluation Criteria

ELIGIBILITY:
* Inclusion Criteria: the standard criteria for treating HCC patients with SBRT : an Eastern Cooperative Oncology Group (ECOG) score of 2, inoperable tumors (e.g. the patient being unfit for surgery, or tumor-related contraindications), and a maximum tumor diameter of 6 cm. The HCC diagnosis could be histological or based on the radiological criteria of the American Association for the Study of Liver Diseases (AASLD)
* Exclusion Criteria:no follow-up by MR imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients records were extracted from the electronic health record system of Institut de Cancérologie de Lorraine
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2013-04-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
tumor response assessments | Within the 24 months after SBRT
  The tumor response was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1